CLINICAL TRIAL: NCT00725790
Title: Multi-Centre, Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Vardenafil in Men With Erectile Dysfunction Caused by Spinal Cord Injury
Brief Title: A Study to Evaluate the Efficacy and Safety of Vardenafil in Men With Erectile Dysfunction Caused by Spinal Cord Injury
Acronym: SCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Rehabilitation Research Center (Other Government)
Responsible Party: Professor Li-Min Liao, China Rehabilitation Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-01
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Spinal Cord Injury
MeSH Terms: conditions — Erectile Dysfunction; Spinal Cord Injuries | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental): Vardenafil treatment group
  Interventions: Drug: Vardenafil
- B (Placebo Comparator): Placebo treatment group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil — 10 mg vardenafil on demand treatment for first 4 weeks.
  A decision is made at week 4 to either maintain the previous dosage regimen or to up-titrate to 20 mg per dose of vardenafil or down-titrate to 5 mg per dose of vardenafil during the subsequent 4 week double-blind treatment period.
  A decision is made at week 8 to either maintain the previous dosage regimen or to up-titrate to 20 mg per dose of vardenafil or down-titrate to 5 mg per dose of vardenafil during the subsequent 4 week double-blind treatment period.
  Arms: A
Drug: Placebo — 10 mg placebo on demand treatment for first 4 weeks.
  A decision is made at week 4 to either maintain the previous dosage regimen or to up-titrate to 20 mg per dose of placebo or down-titrate to 5 mg per dose of placebo during the subsequent 4 week double-blind treatment period.
  A decision is made at week 8 to either maintain the previous dosage regimen or to up-titrate to 20 mg per dose of placebo or down-titrate to 5 mg per dose of placebo during the subsequent 4 week double-blind treatment period.
  Arms: B

SUMMARY:
The purpose of this study is to determine if 12 weeks of flexible-dose vardenafil therapy demonstrates superior efficacy compared to placebo in subjects with ED solely secondary to a traumatic spinal cord injury

DETAILED DESCRIPTION:
According to the Massachusetts Male Aging Study, erectile dysfunction (ED) is estimated as affecting approximately 30 million American men and 100 million men worldwide. The study also reported that approximately 52% of males aged 40-70 experience some degree of ED. Prevalence has been shown to increase with age, with an estimated 40% of the responders experiencing ED at age 40, whereas, 67% had difficulties by age 75.

Considerable advances have been made since the NIH Consensus statement that defined ED as the persistent inability to achieve and maintain an erection sufficient for satisfactory sexual performance. However, one thing remains the same, sexuality continues to be a driving force in our society today. Many men with erectile dysfunction suffer from issues of self esteem, self worth, the creation and maintenance of interpersonal relationships and in general, wrestle with an overall altered sense of wellbeing. Damage to personal relationships can ensue; and the anger, depression, and anxiety engendered spill over into all aspects of life.

VIAGRA(sildenafil), administered as a flexible-dose regimen, has demonstrated to be an effective and well-tolerated treatment for ED in spinal cord injury sufferers.This is a multi-centre, prospective, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of vardenafil in men with erectile dysfunction caused by spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old, had ED more than 6 months
2. Traumatic spinal cord injury was the sole cause of ED
3. Patients had been in a heterosexual relationship for at least 1 month
4. Documented written informed consent.

Exclusion Criteria:

1. Presence of symptomatic active urinary tract infection, indwelling urethral catheter.
2. Patients who have used any kind of PDE-5i prior to the study
3. Other conditions that may cause ED such as history of radical prostatectomy, diabetes mellitus, anatomic penile abnormality and primary hypoactive sexual desire
4. History of symptomatic uncontrolled autonomic dysreflexia; postural hypotension
5. Cardiovascular abnormality such as unstable angina pectoris, myocardial infarction or stroke, electrocardiographic ischemia or life-threatening arrhythmia, resting systolic blood pressure>170 or <90 mmHg, diastolic pressure >110mmHg
6. Retinitis pigmentosa
7. Patients who currently were using any of the following medications: nitrates, nitric oxide donors, androgen or antiandrogen, anticoagulants, trazodone, erythromycin, azole antifungals, other contraindicative medications in package insert
8. Other contraindications in package insert

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
EF domain score of IIEF | week 12

SECONDARY OUTCOMES:
IIEF/SEP/GAQ | at week 4, week 8, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Liao, Dr., Principal Investigator — China Rehabilitation Research Center
Locations (1):
- Beijing Boai Hospital Affiliated to China Rehabilitation Research Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Korenman SG. New insights into erectile dysfunction: a practical approach. Am J Med. 1998 Aug;105(2):135-44. doi: 10.1016/s0002-9343(98)00191-0. PMID 9727821